CLINICAL TRIAL: NCT02244710
Title: EndoTic - Endothelium and Ticagrelor: Pharmacological Effects Beyond Antiplatelet Therapy
Brief Title: EndoTic - Endothelium and Ticagrelor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Investigación Sanitaria en León (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISSBRIL0205; 2013-005042-11 (EudraCT Number)
Record Dates: First submitted 2014-09-11; First posted 2014-09-19 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: Circulating Endothelial Cells; Endothelial Progenitor Cells; Acute coronary syndrome (ACS); Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor (Experimental): 180mg initial dose next day 90mg BID
  Interventions: Drug: Ticagrelor vs Clopidogrel
- Clopidogrel (Active Comparator): 600mg po initial dose and 75mg qd starting next day
  Interventions: Drug: Ticagrelor vs Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor vs Clopidogrel

SUMMARY:
Randomized clinical trial to assess the influence of treatment with ticagrelor or clopidogrel in the number of CECs (Circulating Endothelial Cells) and EPCs (Endothelial Progenitor Cells) in patients with ACS (Acute Coronary Syndrome), from baseline levels to chronic levels (1 month).

DETAILED DESCRIPTION:
ACS Patients in both treatment groups will be assessed:

Baseline, 48h and 1 month cell counts will be done for CECs and EPCs Platelet Function at 48h and 1month Adverse Events, ECG and blood testing result will be also collected

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign Informed Consent Form
* 18 yr or older
* Male and female (post menopause or contraception treatment)
* ACS diagnosed with elevation of myocardial infarction biomarkers (as of 3rd Universal Definition of MI)
* Planned invasive strategy (coronariography performed within 72hrs after admission)

Exclusion Criteria:

* Aspirin, clopidogrel or ticagrelor allergy.
* Hemorrhagic diathesis or very high risk of bleeding.
* Current treatment with oral anticoagulants, thienopyridines or ticagrelor.
* Limited life expectancy.
* Elective surgery planned.
* High chance of not being able to complete the follow-up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of cells | Baseline
  EPC (Endothelial Progenitor Cells) CEC (Circulating Endothelial Cells)
Number of cells | 48 hours after last chest pain episode
  EPC (Endothelial Progenitor Cells) CEC (Circulating Endothelial Cells)
Number of cells | 1 month visit
  EPC (Endothelial Progenitor Cells) CEC (Circulating Endothelial Cells)

SECONDARY OUTCOMES:
Platelet reactivity | At the time of coronary angiography
  As determined by P2Y12 kits, VerifyNow®
Platelet reactivity | 1 month visit
  As determined by P2Y12 kits, VerifyNow®

OTHER OUTCOMES:
Safety: Bleeding and ischemic adverse events | 18 months (Study duration)
  Adverse Events collection

CONTACTS AND LOCATIONS:
Overall Officials: Armando Pérez de Prado, MD, PhD, Principal Investigator — Fundación Investigación Sanitaria en León; M. Belen Vidriales Acosta, MD, PhD, Study Director — University of Salamanca
Locations (3):
- Spain (3):
  - Hospital Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital de Leon, León, Leon
  - Hospital Universitario de Salamanca, Salamanca